CLINICAL TRIAL: NCT02350972
Title: Inducing Systemic Immunity and Regressions in Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Principal Investigator, Fred T. Valentine, Professor of Medicine, NYU Langone Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S-1300774
Record Dates: First submitted 2015-01-14; First posted 2015-01-30 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Metastatic Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Cytokines; Chemokines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous cytokiines (Experimental): Autologous cytokines obtained from patients' blood mononuclear cells injected in volumes of 0.1 ml
  Interventions: Biological: Autologous cytokines

INTERVENTIONS:
Biological: Autologous cytokines — Sterile autologous cytokines were injected weekly into multiple metastatic nodules while other nodules in the patient were never injected and were monitored for the development of dense lymphocytic infiltrates as evidence of an induced immune response.
  Other Names: cytokine/chemokine

SUMMARY:
In patients with multiple metastatic nodules of melanoma, the investigators evaluated whether autologous cytokines injected into cutaneous metastases would induce a systemic immune response as evidenced by the accumulation of dense lymphocytic infiltrates in metastases that had never been injected. Such immune responses were observed, and often the never-injected metastasis regressed completely. 20% of patients remained free of disease for greater than 5 years.

DETAILED DESCRIPTION:
Lymphocytic infiltrates were seen in never-injected nodules only after several weeks of injections elsewhere. No adverse events were seen. The tumor-infiltrating lymphocytes were able to kill autologous melanoma ex vivo. Some patients who experienced complete regressions of all metastases lived without disease for over 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Multiple cutaneous or subcutaneous metastases of melanoma

Exclusion Criteria:

* Visceral metastases on admission.
* No current chemotherapy or immunotherapy.
* Note study performed between 1978 and 2002 before current therapies were available.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 1978-07; Primary Completion 2002-05 (Actual); Study Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
Immune responses as evidenced by lymphocytic infiltrates in never-injected nodules. | Cutaneous nodules were biopsied by a surgeon afer 8 to 20 weeks of injections.
  The biopsies were examined by a licensed pathologist for the presence of dense lymphocytic infiltrates.

SECONDARY OUTCOMES:
Complete regression of a metastasis | Complete regressions of all injected and never-injected metastases occurred in different pts after 13 weeks to 48 months of injections. Pts with progressive disease were switched to chemotherapy at any point in the study.
  70 % of patients had at least one nodule regress. 40 % had all metastases completely regress for 5 to 20 years (median 60 months).

CONTACTS AND LOCATIONS:
Overall Officials: Fred T. Valentine, M.D., Principal Investigator — NYU Langone Health